CLINICAL TRIAL: NCT01331083
Title: A Phase II Study of PX-866 in Patients With Recurrent or Metastatic Castration Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Oncothyreon Canada Inc. (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I205
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PX-866

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PX-866 (Experimental)
  Interventions: Drug: PX-866

INTERVENTIONS:
Drug: PX-866 — PX-866: 8mg orally taken daily

SUMMARY:
The purpose of this study is to find out whether the new drug PX-866 will slow the growth of your prostate cancer. The investigators will also watch you carefully for any side effects that PX-866 might cause.

DETAILED DESCRIPTION:
PX 866 is a new type of drug that inhibits a molecule related to cancer cell growth. While this molecule is also found in normal cells, it is much more active in some cancer cells, so inhibiting the molecule with PX-866 is hoped to slow the growth of cancer cells. Laboratory tests show that it may help slow the growth of prostate cancer in animals, but it is not known whether it will have the same effects in humans. PX-866 has been studied in some cancer patients to find out safe doses that can be given but it has not undergone study in prostate cancer. This study will be the first study of PX-866 in prostate cancer.

Health Canada has not approved the sale or use of PX-866 to treat prostate cancer, although they have approved its use in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or cytological diagnosis of adenocarcinoma of the prostate.
* All patients must have formalin fixed paraffin embedded tissue (from their primary or metastatic tumour) available for translational studies.
* Presence of clinically and/or radiologically documented disease (measureable or non-measurable). All radiology studies must be performed within 28 days prior to registration (within 35 days if negative).
* Androgen ablation must include either medical or surgical castration. If the patient is receiving medical androgen ablation, a castrate level of testosterone (< 1.7 nmol/L) must be present.
* Patients must have metastatic or locally recurrent disease, for which no curative therapy exists and for which systemic therapy is indicated.
* No prior chemotherapy regimens for recurrent disease

For Part A, patients must have progression defined as:

PSA Progression: A rising PSA, while receiving androgen ablative therapy, with 2 subsequent rises over a reference value (not necessarily consecutively), measured a minimum of one week apart. The PSA that confirms progression must have a value of ≥ 5 ng/ml and must be performed no longer than 7 days prior to trial registration.

OR Radiological Progression: defined as the development of new metastatic lesions with a stable or rising PSA.

Patients entered to Part B of the study (after 2nd stage of accrual completed) must have a rise in their PSA while on abiraterone/prednisone continuing at time of registration (≥ 25% higher from baseline or nadir, whichever is lowest).

* The PSA must be ≥5 ng/ml at the time of study entry.
* ECOG performance of 0, 1 or 2.
* Age ≥ 18 years of age.

Previous therapy:

Surgery:

Previous major surgery is permitted provided that it has been at least 14 days prior to patient registration and that wound healing has occurred.

Hormonal Therapy:

Prior hormone therapy is required. Patients must be hormone refractory and have discontinued anti-androgens for at least 4 weeks prior to study entry (at least 6 weeks for bicalutamide). Therapy with LHRH agonist must continue for those prostate cancer patients already receiving this treatment at the time of enrollment. If the patient has discontinued the LHRH agonist, this must be restarted (if not surgically castrated) and the castrate level of testosterone must be present. Prior therapy with CYP17 inhibitors (e.g. abiraterone, ketoconazole) or novel anti-androgens (e.g. MDV3100) is permitted.

Part B: Patients must be hormone refractory and have discontinued anti-androgens for at least 4 weeks prior to study entry (at least 6 weeks for bicalutamide). Therapy with LHRH agonist must continue for those prostate cancer patients already receiving this treatment at the time of enrollment. If the patient has discontinued the LHRH agonist, this must be restarted (if not surgically castrated) and the castrate level of testosterone must be present. All patients must currently be receiving abiraterone.

Radiation:

Prior external beam radiation is permitted provided a minimum of 2 weeks has elapsed between the last dose and enrollment to the trial. Exceptions may be made for low dose, non-myelosuppressive radiotherapy after consultation with NCIC CTG. Prior strontium is not permitted.

- Laboratory Requirements (must be done within 7 days prior to registration)

Hematology:

Granulocytes (AGC) ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L

Biochemistry:

Serum creatinine ≤ 1.5 x UNL Total bilirubin ≤ 1.5 x UNL ALT and AST ≤ 1.5 x UNL Glucose ≤ 8.9 mmol/L (≤ Grade 1) PSA ≥ 5ng/mL

-Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration.

Exclusion Criteria:

* Patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer or solid tumours curatively treated with no evidence of disease for >=3 years.
* Known HIV-positive patients.
* Uncontrolled diabetes mellitus.
* Patients with upper gastrointestinal or other conditions that would preclude compliance or absorption of oral medication are not eligible.
* Patients with active or uncontrolled infections, or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Patients with history of central nervous system metastases or untreated spinal cord compression.
* Patients who have had prior treatment with a PI3 kinase inhibitor.
* Men who are not sterile unless they use an adequate method of birth control.
* Patients enrolled to Part B must be suitable for continued therapy with abiraterone/prednisone.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-09-09 (Actual); Primary Completion 2015-01-13 (Actual); Study Completion 2015-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, Study Chair — BCCA Vancouver Cancer Centr; Sebastien Hotte, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences
Locations (10):
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hotte SJ, Chi KN, Joshua AM, Tu D, Macfarlane RJ, Gregg RW, Ruether JD, Basappa NS, Finch D, Salim M, Winquist EW, Torri V, North S, Kollmannsberger C, Ellard SL, Eigl BJ, Tinker A, Allan AL, Beja K, Annala M, Powers J, Wyatt AW, Seymour L; Canadian Cancer Trials Group (formerly NCIC Clinical Trials Group). A Phase II Study of PX-866 in Patients With Recurrent or Metastatic Castration-resistant Prostate Cancer: Canadian Cancer Trials Group Study IND205. Clin Genitourin Cancer. 2019 Jun;17(3):201-208.e1. doi: 10.1016/j.clgc.2019.03.005. Epub 2019 Mar 15. PMID 31056399

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Patients with castration resistant prostate cancer, who have received no prior chemotherapy regimens for recurrent disease, treated by PX-866 at 8mg when given orally daily
- Group B: Patients with castration resistant prostate cancer, who have had PSA progression while receiving abiraterone/prednisonee, treated by PX-866 at 8mg when given orally daily
Period: Overall Study
Arm/Group | Group A | Group B
Started | 43 | 25
Completed | 43 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in this study
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 43 | 25 | 68
Age, Continuous [Median (Full Range); unit: years] | 70 [51 to 90] | 72 [52 to 84] | 71 [51 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 25 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 25 | 68
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 43 | 25 | 68

OUTCOME MEASURES:

1. Primary Outcome: Lack of Disease Progression at 12 Weeks
Description: Proportion of patients without evidence of progression (objective progression, defined as an increase in sum of diameters of target lesions of at least 20% above the lowest (or baseline) value (minimum of 5 mm increase) OR the appearance of unequivocal increase in non-measurable/non-target disease OR the appearance of new lesions, or PSA progression, defined as a rise in PSA of 25% (minimum 5 ng/ml) above baseline value or nadir, whichever is lowest, and confirmed by a second increasing value at least 3 weeks later) at 12 weeks after start of therapy
Time Frame: 12 weeks
Population: All patients enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 25
Participants | 14 | 11

2. Secondary Outcome: PSA Response Rate
Description: Proportion of patients with PSA response defined as a > 50% fall in PSA (minimum of 5 ng/ml) from baseline maintained for > 4 weeks without evidence of disease progression otherwise
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 25
Participants | 1 | 0

3. Secondary Outcome: Objective Response Rate
Description: Proportion of patients with objective response defined as 30% decrease in the sum of the longest diameters of the target lesions (partial response) maintained for at least 4 weeks, or complete disappearance of disease and cancer related symptoms (complete response), also maintained for at least 4 weeks
Time Frame: 12 weeks
Population: All patients enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 43 | 25
Participants | 2 | 0

4. Secondary Outcome: Change in Circulating Tumour Cell Number During Treatment
Description: Proportion of patients with Favorable circulating tumour cell (CTC) conversion (< 5 CTC/7.5 mL)
Time Frame: 12 weeks
Population: All patients with CTC assessed (not required for Group B patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 25 | 0
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 6/43 | 5/25
Serious Adverse Events (participants affected / at risk) | 8/43 | 5/25
Other Adverse Events (participants affected / at risk) | 43/43 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=43) | Group B (N=25)
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Lung infection (Infections and infestations) | 2 | 0
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hematuria (Renal and urinary disorders) | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Esophageal obstruction (Gastrointestinal disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Fever (General disorders) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Pain (General disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=43) | Group B (N=25)
Abdominal pain (Gastrointestinal disorders) | 8 | 4
Watering eyes (Eye disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 19 | 14
Diarrhea (Gastrointestinal disorders) | 31 | 18
Dyspepsia (Gastrointestinal disorders) | 9 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 33 | 13
Vomiting (Gastrointestinal disorders) | 14 | 11
Chills (General disorders) | 3 | 1
Edema limbs (General disorders) | 8 | 6
Fatigue (General disorders) | 30 | 21
Fever (General disorders) | 3 | 3
Pain (General disorders) | 14 | 3
Other infections and infestations (Infections and infestations) | 6 | 1
Anorexia (Metabolism and nutrition disorders) | 21 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 6
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 4 | 0
Dizziness (Nervous system disorders) | 4 | 4
Dysgeusia (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 10 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 10 | 3
Anxiety (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 8 | 2
Hematuria (Renal and urinary disorders) | 5 | 2
Urinary frequency (Renal and urinary disorders) | 16 | 6
Urinary retention (Renal and urinary disorders) | 3 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 8 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1
Hot flashes (Vascular disorders) | 10 | 7
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 4
Other gastrointestinal disorders (Gastrointestinal disorders) | 1 | 5
Bruising (Injury, poisoning and procedural complications) | 1 | 3
Weight loss (Investigations) | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 2 | 3
Urinary urgency (Renal and urinary disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No